CLINICAL TRIAL: NCT00147940
Title: Correlation of Nasal Volume and Cross-Sectional Area With Nasalance Scores as Measured by Acoustic Rhinometry and Nasometry
Brief Title: Correlation of Nasal Volume, Cross-Sectional Area With Nasalance Scores Measured by Acoustic Rhinometry and Nasometry
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13093A
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Allergy
Keywords: Allergy
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Procedure: Acoustic rhinometry (procedure)

SUMMARY:
The purpose of our study is to correlate nasal volume and cross-sectional area with nasalance scores. We will measure nasal volume and cross-sectional area with acoustic rhinometry. Nasalance scores will be determined by Nasometry.

Acoustic rhinometry is a means to study the volume and cross-sectional areas of the nasal cavity in a non-invasive, rapid, convenient and reliable manner. Acoustic rhinometry has the unique advantage of being completely non-invasive, and thus is able to measure nasal patency without the confounding effects of probes or invasive monitoring.

Nasometry is a technique to measure the oral and nasal components of nasalance. Nasalance is the objective measure of the nasal component of speech that is determined by the ratio of sound pressure emitted from the nasal and oral cavities during speech. Nasality is the term used to characterize the nasal component of speech, and is a subjective measure.

Eleven healthy subjects underwent acoustic rhinometry pre and post decongestion using oxymetazoline 0.05% nasal spray. Nasalance scores were based on the readings of three passages: rainbow, zoo, and nasal.

DETAILED DESCRIPTION:
Acoustic rhinometry is a technique that utilizes sound waves to measure nasal patency. The reflections of the waves off of the nasal structures allow one to assess the volume and cross sectional area of the nasal cavity. It is a non-invasive procedure that can be performed in a rapid, convenient, and reliable manner. There is minimal discomfort for the patient and it can be performed easily in the office. There is no distortion of nasal anatomy or functioning as a result of the procedure.

Nasometry is a technique to measure the oral and nasal components of nasalance. Nasalance is an objective measure of the nasal component of speech that is determined by the ratio of acoustic pressures emitted from the nasal and oral cavities. 'Nasality' is the term used to characterize the nasal component of speech, and is a subjective measure.

The Nasometer (Kay Elemetrics Corp Lincoln Park, NJ) is a computer-based device that analyzes acoustic energy that is emitted from the oral and the nasal cavity during speech. It consists of two microphones that are separated by a plate. The upper microphone measures nasally emitted acoustic energy, and the lower microphone measure the acoustic energy emitted from the oral cavity.

Nasalance is an important measure in speech pathology. In situations where velopharyngeal competence is in question, nasometry objectively documents the nasal component of speech as normal, hypemasal or hyponasal. It has been found to be of tremendous benefit in the management of patients with cleft palate and velopharyngeal incompetence. The subject is relaxed, and is fitted with a headgear apparatus. This apparatus is placed such that a plate lies in a horizontal plane that rests midway between the nose and the mouth. There are microphones on the upper and lower surfaces of the plate that capture sound energy produced from the nasal and oral cavities respectively. The subject is then asked to read standard passages. The three most commonly used passages are described here, and will be used in our study. The 'Rainbow' passage is most representative of standard English speech. The 'Zoo' passage has no nasal consonants, and the 'Nasal' passage has the highest number of nasal consonants.

While the subject is reading, the microphone captures sound pressure levels which are emitted from the nasal and the oral cavities. This data is analyzed by the attached computer and presented graphically. The computer also provides a nasalance score for each of three above- mentioned passages. Normative data is available for each of these passages for adults and children. By comparing the data obtained from the subject with the normative means and standard deviations, the investigator can categorize the subject's voice as normal, hyponasal or hypernasal. The nasalance score that is generated can also be used to monitor the efficacy of speech therapy and surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over the age of 18 years who no gross nasal deformity

Exclusion Criteria:

* Pregnant or nursing females
* Subjects younger than 18 years
* Allergy to the drug oxymetazoline
* Inability to read a simple standard English passage
* History of heart disease, hypertension, renal, liver or lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08

PRIMARY OUTCOMES:
Nasal volume

SECONDARY OUTCOMES:
Nasalance scores

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Martin, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Moinuddin R, Mamikoglu B, Barkatullah S, Corey JP. Detection of the nasal cycle. Am J Rhinol. 2001 Jan-Feb;15(1):35-9. doi: 10.2500/105065801781329473. PMID 11258653
- [Background] Corey JP, Houser SM, Ng BA. Nasal congestion: a review of its etiology, evaluation, and treatment. Ear Nose Throat J. 2000 Sep;79(9):690-3, 696, 698 passim. PMID 11011488
- [Background] Corey JP, Nalbone VP, Ng BA. Anatomic correlates of acoustic rhinometry as measured by rigid nasal endoscopy. Otolaryngol Head Neck Surg. 1999 Nov;121(5):572-6. doi: 10.1016/S0194-5998(99)70058-6. PMID 10547472
- [Background] Mamikoglu B, Houser S, Akbar I, Ng B, Corey JP. Acoustic rhinometry and computed tomography scans for the diagnosis of nasal septal deviation, with clinical correlation. Otolaryngol Head Neck Surg. 2000 Jul;123(1 Pt 1):61-8. doi: 10.1067/mhn.2000.105255. PMID 10889483
- [Background] Corey JP, Gungor A, Nelson R, Fredberg J, Lai V. A comparison of the nasal cross-sectional areas and volumes obtained with acoustic rhinometry and magnetic resonance imaging. Otolaryngol Head Neck Surg. 1997 Oct;117(4):349-54. doi: 10.1016/S0194-5998(97)70125-6. PMID 9339795
- [Background] Seaver EJ, Dalston RM, Leeper HA, Adams LE. A study of nasometric values for normal nasal resonance. J Speech Hear Res. 1991 Aug;34(4):715-21. doi: 10.1044/jshr.3404.715. PMID 1956179
- [Background] Williams RG, Eccles R, Hutchings H. The relationship between nasalance and nasal resistance to airflow. Acta Otolaryngol. 1990 Nov-Dec;110(5-6):443-9. doi: 10.3109/00016489009107467. PMID 1704676
- [Background] Mayo R, Floyd LA, Warren DW, Dalston RM, Mayo CM. Nasalance and nasal area values: cross-racial study. Cleft Palate Craniofac J. 1996 Mar;33(2):143-9. doi: 10.1597/1545-1569_1996_033_0143_nanavc_2.3.co_2. PMID 8695622
- [Background] Dalston RM, Warren DW, Dalston ET. A preliminary investigation concerning the use of nasometry in identifying patients with hyponasality and/or nasal airway impairment. J Speech Hear Res. 1991 Feb;34(1):11-8. doi: 10.1044/jshr.3401.11. PMID 2008065